CLINICAL TRIAL: NCT01832103
Title: A Phase I Study to Evaluate the Pharmacokinetics of MK-7145 Following Single Dose Administration in Patients With Moderate Renal Insufficiency
Brief Title: The Pharmacokinetics of MK-7145 Following Single Dose Administration in Participants With Moderate Renal Insufficiency (MK-7145-018)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7145-018; 2013-000838-35 (EudraCT Number)
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — MK-7145

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK-7145 (Experimental): MK-7145 2 mg IR administered as a single oral dose.
  Interventions: Drug: MK-7145

INTERVENTIONS:
Drug: MK-7145

SUMMARY:
The primary purpose of this study is to obtain a preliminary pharmacokinetic profile of MK-7145 2 mg immediate release (IR) following single-dose administration in male participants with moderate renal insufficiency. In addition, the study will evaluate the pharmacodynamic effect of a single dose of MK-7145 2 mg IR on 24-hour net natriuresis in male participants with moderate renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18 to 35 kg/m^2
* Nonsmoker and/or have not used nicotine or nicotine-containing products

for at least 3 months prior to enrollment

* Estimated glomerular filtration rate (eGFR) 30 to 60 mL/min/1.73 m^2

Exclusion Criteria:

* History of stroke, chronic seizures, or major neurological disorder
* Ongoing, clinically significant endocrine, gastrointestinal, cardiovascular,

hematological, hepatic, immunological, respiratory, or genitourinary abnormalities or diseases

* Systolic blood pressure (SBP) ≤95 mmHg or >160 mmHg, or diastolic blood

pressure (DBP) ≤45 mmHg or >95 mmHg

* History of neoplastic disease except for adequately treated non-melanomatous skin carcinoma
* Unable to refrain from, or anticipates the use of, strong/moderate cytochrome P450 3A4 (CYP3A4) inhibitors
* Consumes excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages, wine, or distilled spirits per day
* Consumes excessive amounts of caffeine, defined as greater than 6 servings of coffee, tea, cola, or other caffeinated beverages per day
* Had major surgery or donated blood within 8 weeks prior to enrollment
* Has participated in another investigational study within 4 weeks prior
* History of significant multiple and/or severe allergies (including latex allergy), or has had an anaphylactic reaction or significant intolerance to prescription or nonprescription drugs or food
* Currently a regular user of illicit drugs, or has a history of drug (including alcohol) abuse within approximately 6 months
* Has active or has a history of nephrolithiasis
* Has had a kidney removed or has a functioning renal transplant

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma-Time Curve From 0 to Infinity (AUC0-∞) of MK-7145 2 mg IR Following Single Dose Administration | Up to 48 Hours Post Dose
Maximum Plasma Concentration (Cmax) of MK-7145 2 mg IR Following Single Dose Administration | Up to 48 Hours Post Dose
Time to Maximum Plasma Concentration (Tmax) of MK-7145 2 mg IR Following Single Dose Administration | Up to 48 Hours Post Dose
Apparent Half-Life (t 1/2) of MK-7145 2 mg IR Following Single Dose Administration | Up to 48 Hours Post Dose
Oral Clearance (CL/F) of MK-7145 2 mg IR Following Single Dose Administration | Up to 24 Hours Post Dose
Oral Volume of Distribution (V/F) of MK-7145 2 mg IR Following Single Dose Administration | Up to 48 Hours Post Dose

SECONDARY OUTCOMES:
Change From Baseline in 24-Hr Urine Natriuresis (UNa0-24) | 24 Hours Prior to Dosing (Baseline) and Up to 24 Hours Post Dose